CLINICAL TRIAL: NCT04704921
Title: A Randomized, Partially Masked, Controlled, Phase 2b/3 Clinical Study to Evaluate the Efficacy and Safety of RGX-314 Gene Therapy in Participants With nAMD (ATMOSPHERE)
Brief Title: Pivotal 1 Study of ABBV-RGX-314 (Also Known as RGX-314) Gene Therapy Administered Via Subretinal Delivery One Time in Participants With nAMD
Acronym: ATMOSPHERE
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: REGENXBIO Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RGX-314-2104; M23-416 (Other: AbbVie Inc)
Record Dates: First submitted 2021-01-08; First posted 2021-01-12 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: AMD; nAMD; Wet Age-related Macular Degeneration; wAMD; Wet AMD; CNV; Neovascular AMD; Neovascular Age-related Macular Degeneration; Choroidal Neovascularization
Keywords: Age-Related Macular Degeneration; Neovascular Age-Related Macular Degeneration; Macular Degeneration; Wet Macular Degeneration; Choroidal Neovascularization; Retinal Degeneration; Retinal Diseases; Eye Diseases; Ranibizumab; Angiogenesis Inhibitors; Angiogenesis Modulating Agents; Growth Substances; Physiological Effects of Drugs; Growth Inhibitors; Antineoplastic Agents; Gene therapy; Anti-vascular endothelial grown factory therapy; Anti-VEGF therapy
MeSH Terms: conditions — Choroidal Neovascularization; Macular Degeneration; Wet Macular Degeneration; Retinal Degeneration; Retinal Diseases; Eye Diseases | interventions — Ranibizumab

STUDY DESIGN:
Intervention Model Description: 2 ABBV-RGX-314 treatment arms, 1 control arm (ranibizumab)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The administration of ABBV-RGX-314 requires an outpatient surgical procedure performed in an operating room, while the active control, ranibizumab, is administered via intravitreal injection in an office setting. This study will be partially masked which will include masking of key study assessors and study drug dose.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- ABBV-RGX-314 Dose 1 (Experimental): ABBV-RGX-314 Dose 1 administered via subretinal delivery one time.
  Interventions: Genetic: ABBV-RGX-314
- ABBV-RGX-314 Dose 2 (Experimental): ABBV-RGX-314 Dose 2 administered via subretinal delivery one time.
  Interventions: Genetic: ABBV-RGX-314
- Control Arm (Active Comparator): Ranibizumab administered via intravitreal injection approximately every 28 days
  Interventions: Biological: Ranibizumab (LUCENTIS®)

INTERVENTIONS:
Genetic: ABBV-RGX-314 — AAV8 vector containing a transgene for anti-VEGF Fab (Dose 1)
  Other Names: surabgene lomparvovec; RGX-314
  Arms: ABBV-RGX-314 Dose 1
Genetic: ABBV-RGX-314 — AAV8 vector containing a transgene for anti-VEGF Fab (Dose 2)
  Other Names: surabgene lomparvovec; RGX-314
  Arms: ABBV-RGX-314 Dose 2
Biological: Ranibizumab (LUCENTIS®) — 0.5 mg (0.05 mL of 10 mg/mL solution) administered by intravitreal injection approximately every 28 days
  Other Names: Ranibizumab (anti-VEGF agent)
  Arms: Control Arm

SUMMARY:
ABBV-RGX-314 (also known as RGX-314) is being developed as a novel one-time gene therapy for the treatment of neovascular (wet) age-related macular degeneration (wet AMD or nAMD). Wet AMD is characterized by loss of vision due to new, leaky blood vessel formation in the retina. Wet AMD is a significant cause of vision loss in the United States, Europe and Japan, with up to 2 million people living with wet AMD in these geographies alone. Current anti-vascular endothelial growth factor (anti-VEGF) therapies have significantly changed the landscape for treatment of wet AMD, becoming the standard of care due to their ability to maintain or prevent progression of vision loss in the majority of patients. These therapies, however, require life-long intraocular injections, typically repeated every 4 to 16 weeks in frequency, to maintain efficacy. Due to the burden of these treatments, patients often experience a decline in vision with reduced frequency of treatment over time.

DETAILED DESCRIPTION:
This randomized, partially masked, active-controlled, Phase 2b/3 clinical study will evaluate the efficacy and safety of ABBV-RGX-314 gene therapy in participants with nAMD. The study will evaluate 2 dose levels of ABBV-RGX-314 relative to an active comparator. The primary endpoint of this study is the mean change from baseline in best-corrected visual acuity (BCVA) of ABBV-RGX-314 relative to ranibizumab at Week 54. Approximately 630 participants who meet the inclusion/exclusion criteria, will be enrolled into one of 3 arms.

A bilateral treatment substudy conducted at US sites is an open-label, partially randomized, parallel arm study to evaluate the safety and efficacy of subretinal ABBV-RGX-314 administered bilaterally in participants who have bilateral nAMD. Previously treated crossover participants from the control arm of the main study who crossed over and received ABBV-RGX-314 in the study eye will receive the same ABBV-RGX-314 dose in the contralateral eye (ie, same dose as in the study eye), and newcomers (participants who have not been randomized in an ABBV-RGX-314 study) and untreated crossover participants (ongoing control participants in the main study who have completed Week 54 but have not crossed over to receive ABBV-RGX-314 in the main study) will be randomized in a 2:1 ratio to receive ABBV-RGX-314 Dose 1 or ABBV-RGX-314 Dose 2 in both eyes. Up to 15 participants who qualify for the substudy will be enrolled and followed for a minimum of 50 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 50 years and ≤ 89 years
2. An ETDRS BCVA letter score between ≤ 78 and ≥ 40 in the study eye
3. Diagnosis of subfoveal CNV secondary to AMD in the study eye previously treated with anti-VEGF
4. Must be pseudophakic (at least 12 weeks postcataract surgery) in the study eye.
5. Willing and able to provide written, signed informed consent for this study
6. Participants must have demonstrated a meaningful response to anti-VEGF therapy at study entry

Inclusion Criteria (Bilateral Treatment Substudy)*:

1. An ETDRS BCVA letter score between ≤ 83 and ≥ 40 in both eyes
2. Diagnosis of subfoveal choroidal neovascularization (CNV) secondary to AMD in both eyes
3. Must be pseudophakic (at least 12 weeks postcataract surgery) in both eyes
4. Willing and able to provide written, signed informed consent for this study
5. Newcomers must have active disease in the study eye; crossover participants must have active disease in the eye not treated in the main study

Exclusion Criteria:

1. CNV or macular edema in the study eye secondary to any causes other than AMD
2. Subfoveal fibrosis or atrophy in the study eye, as determined by CRC
3. Any condition in the investigator's opinion that could limit VA improvement in the study eye
4. Active or history of retinal detachment, or current retinal tear that cannot be treated, in the study eye
5. Advanced glaucoma or history of secondary glaucoma in the study eye
6. History of intraocular surgery in the study eye within 12 weeks prior to randomization
7. History of intravitreal therapy in the study eye, such as intravitreal steroid injection or investigational product, other than anti-VEGF therapy, in the 6 months prior to Screening Visit 1
8. Prior treatment with gene therapy
9. Recent myocardial infarction, cerebrovascular accident, or transient ischemic attack within the past 6 months

Exclusion Criteria (Bilateral Treatment Substudy)*:

1. CNV or macular edema in either eye secondary to any causes other than AMD
2. Subfoveal fibrosis or atrophy in either eye
3. Any condition in the investigator's opinion that could limit VA improvement in either eye
4. Active or history of retinal detachment, or current retinal tear that cannot be treated in either eye
5. Advanced glaucoma or history of secondary glaucoma in either eye
6. Myocardial infarction, cerebrovascular accident, or transient ischemic attack within the past 6 months
7. History of intraocular surgery in either eye within 12 weeks prior to randomization
8. History of intravitreal therapy in either eye, such as intravitreal steroid injection or investigational product, other than anti-VEGF therapy, in the 6 months prior to screening
9. Prior treatment with gene therapy (*) For previously treated crossover participants, criteria apply to the eye not treated in the main study only.

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 630 (Estimated)
Dates: Start 2020-12-29 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in Best Corrected Visual Acuity (BCVA) | At Week 54
  BCVA measured by Early Treatment Diabetic Retinopathy Study (ETDRS)
Bilateral Treatment Substudy: Incidence of ocular AEs and any SAEs | Week 50
  Incidence of ocular AEs and any SAEs

SECONDARY OUTCOMES:
Proportion of participants with ≤ 2 supplemental anti-VEGF injections through Week 54 (ABBV-RGX-314 randomized participants) | Through Week 54
  Proportion of supplemental anti-VEGF injections.
Proportion of participants with no supplemental anti-VEGF injections through Week 54 (ABBV-RGX-314 randomized participants) | Through Week 54
  Proportion of supplemental anti-VEGF injections.
Incidences of ocular and overall AEs over 54 weeks | Through Week 54
  AEs over 54 weeks
Incidences of ocular and overall AEs over 98 weeks | Through Week 98
  AEs over 98 weeks
Mean change from baseline in BCVA to Week 98 (ABBV-RGX-314 randomized participants) based on the ETDRS score | Week 98
  BCVA measured by ETDRS
Proportion of participants with worsened BCVA | Week 54; Week 98
  Proportion with worsened BCVA
Proportion of participants with improved BCVA | Week 54; Week 98
  Proportion with improved BCVA
Proportion of participants (1) gaining > 0 letters; (2) losing > 0 letters; maintaining vision (not losing ≥ 15 letters) compared with baseline as per BCVA | Week 54; Week 98
  Proportion gaining or losing > 0 letters based on ETDRS score; proportion maintaining vision
Mean change from baseline in BCVA for participants who received 0 or more supplemental anti-VEGF injections (ABBV-RGX-314 randomized participants) | Week 54
  Mean change in BCVA based on ETDRS score for participants who received 0 or more supplemental anti-VEGF injection
Mean change from Week 54 to Week 98 in BCVA (control arm participants who cross over to ABBV-RGX-314) | Week 54 to Week 98
  Mean change in BCVA based on ETDRS score
Mean change from baseline in CRT as measured by SD-OCT | Week 54; (ABBV-RGX-314 randomized participants) Week 98
  Mean change in CRT as measured by SD-OCT
Mean change from Week 54 to Week 98 in CRT as measured by SD-OCT (control arm participants who cross over to ABBV-RGX-314) | from Week 54 to Week 98
  Mean change in CRT as measured by SD-OCT
Mean change from baseline in CPT as measured by SD-OCT | Week 54; (ABBV-RGX-314 randomized participants) Week 98
  Mean change in CPT as measured by SD-OCT
Mean change from Week 54 to Week 98 in CPT as measured by SD-OCT (control arm participants who cross over to ABBV-RGX-314) | from Week 54 to Week 98
  Mean change in CPT as measured by SD-OCT
Proportion of participants with a reduction in anti-VEGF injection annualized rate through Week 54 and Week 98 compared with the prior year (ABBV-RGX-314 randomized participants) | Through Week 54 and Week 98
  Proportion of participants with a reduction of in anti-VEGF injection annualized rate compared with the prior year
Percent reduction in anti-VEGF injection annualized rate compared with the prior year (ABBV-RGX-314 randomized participants) | Through Week 54 and Week 98
  Supplemental anti-VEGF injection annualized rate
Supplemental anti-VEGF injection annualized rate in the ABBV-RGX-314 arms through Week 54 and Week 98 | Through Week 54 and Week 98
  Supplemental anti-VEGF injection annualized rate
Percent reduction in anti-VEGF injection annualized rate after Week 58 through Week 98 relative to the year prior to the study (control arm participants who cross over to ABBV-RGX-314) | After Week 58 through Week 98
  Percent reduction in anti-VEGF injection annualized rate
Supplemental anti-VEGF injection annualized rate after Week 58 through Week 98 (control arm participants who cross over to ABBV-RGX-314) | After Week 58 to Week 98
  Supplemental anti-VEGF injection annualized rate
22. Time to first supplemental anti-VEGF injection after the Week 2 injection in the ABBV-RGX-314 arms | Week 98
  Time to first supplemental anti-VEGF injection
Time to first supplemental anti-VEGF injection after the Week 58 injection in the control arm participants who cross over to ABBV-RGX-314 | After Week 58 to Week 98
  Time to first supplemental anti-VEGF injection
Mean change from baseline in NEI-VFQ-25 (composite score) at Week 54 and (for ABBV-RGX-314 randomized participants and control arm participants who cross over to ABBV-RGX-314) Week 98 | Week 54; Week 98
  Mean change in NEI VGQ-25 (composite score) at week 54 (control arm participants who cross over to ABBV-RGX-314)
Mean change from baseline in MacTSQ (composite score) at Week 54 and (for ABBV-RGX-314 randomized participants and control arm participants who cross over to ABBV-RGX-314) Week 98 | Week 54; Week 98
  Mean change from baseline in MacTSQ (composite score) at week 54 and (control arm participants who cross over to ABBV-RGX-314) at Week 98
Aqueous ABBV-RGX-314 TP concentrations (ABBV-RGX-314 randomized participants) | Wk -2, Wk 14, Wk 26, Wk 38, Wk 54, and Wk 98
  Aqueous ABBV-RGX-314 TP concentration
Aqueous ABBV-RGX-314 TP concentrations (control arm participants who cross over to ABBV-RGX-314) | Wk 54, Wk 66, Wk 78, Wk 90, and Wk 98
  Aqueous ABBV-RGX-314 TP concentration
Immunogenicity measurements (ABBV-RGX-314 randomized participants) | Wk -2, Wk 14, Wk 26, Wk 38, Wk 54, and Wk 98
  Immunogenicity measurements (serum antibodies to AAV8 and serum antibodies to ABBV-RGX-314 TP)
Immunogenicity measurements (control arm participants who cross over to ABBV-RGX-314) | Wk 54, Wk 66, Wk 78, Wk 90, and Wk 98
  Immunogenicity measurements (serum antibodies to AAV8 and serum antibodies to ABBV-RGX-314 TP)
Bilateral Treatment Substudy: Incidence of nonocular AEs and any AEs of special interest | Week 50
  Nonocular AEs and AEs of Special interest
Bilateral Treatment Substudy: Mean change from Baseline in BCVA at assessed timepoints | Through Week 50
  BCVA measured by ETDRS
Bilateral Treatment Substudy: Mean change from Baseline in CRT at assessed timepoints | Through Week 50
  Mean change in CRT as measured by SD-OCT
Bilateral Treatment Substudy: Supplemental anti-VEGF injection annualized rate | Through Week 50
  Supplemental anti-VEGF injection annualized rate
Bilateral Treatement Substudy: Mean number of supplemental anti-VEGF injections | Through Week 50
  Mean supplemental anti-VEGF injections
Bilateral Treatment Substudy: Proportion of participants with no supplemental anti-VEGF injections | Through Week 50
  Proportion of participants with no supplemental anti-VEGF injections
Bilateral Treatment Substudy: Proportion of particpants with ≤2 supplemental anti-VEGF injections | Through Week 50
  Proportion of participants with ≤2 supplemental anti-VEGF injections
Bilateral Treatment Substudy: Aqueous humor and serum ABBV-RGX-314 TP concentrations | Wk 26, Wk 34, Wk 50
  Aqueous humor and serum ABBV-RGX-314 TP Concentrations
Bilateral Treatment Substudy: Immunogenicity measurements (serum anti-ABBV-RGX-314 TP antibodies, serum anti-AAV8 antibodies) and enzyme-linked immunospot at assessed time points | Wk 18, Wk 34, Wk 50
  Immunogenicity measurements

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (89):
- United States (89):
  - Retinal Research Institute /ID# 256019, Phoenix, Arizona
  - Barnet Dulaney Perkins Eye Center - Sun City /ID# 256055, Sun City, Arizona
  - University of Arkansas for Medical Sciences /ID# 271290, Little Rock, Arkansas
  - Retina Vitreous Assoc Med Grp /ID# 256299, Beverly Hills, California
  - Retinal Diagnostic Center /ID# 256137, Campbell, California
  - The Retina Partners - Encino /ID# 256054, Encino, California
  - Retina Consultants of Orange County /ID# 256152, Fullerton, California
  - Salehi Retina Institute /ID# 263485, Huntington Beach, California
  - UC Irvine/Gavin Herbert Eye Institute /ID# 256145, Irvine, California
  - Northern California Retina Vitreous Associates Medical Group, Inc /ID# 256298, Mountain View, California
  - UCLA Doheny Eye Center /ID# 256120, Pasadena, California
  - California Eye Specialists Medical Group Inc. /ID# 256079, Pasadena, California
  - Retina Consultants of San Diego /ID# 256021, Poway, California
  - Retinal Consultants Medical Group /ID# 256047, Sacramento, California
  - West Coast Retina /ID# 256448, San Francisco, California
  - University of California, San Francisco /ID# 256130, San Francisco, California
  - Orange County Retina Medical Group /ID# 256073, Santa Ana, California
  - California Retina Consultants - Santa Barbara /ID# 256017, Santa Barbara, California
  - Retina Consultants of Southern Colorado /ID# 256069, Colorado Springs, Colorado
  - Southwest Retina Research Center /ID# 256136, Durango, Colorado
  - Colorado Retina Associates /ID# 256121, Lakewood, Colorado
  - Retina Group of New England - Waterford /ID# 256071, Waterford, Connecticut
  - Advanced Research, LLC /ID# 275451, Deerfield Beach, Florida
  - Vitreoretinal Associates, P.A. /ID# 256150, Gainesville, Florida
  - Florida Retina Consultants /ID# 265661, Lakeland, Florida
  - Bascom Palmer Eye Institute - University of Miami /ID# 256072, Miami, Florida
  - Retina Specialty Institute /ID# 256153, Pensacola, Florida
  - Retina Vitreous Associates of Florida - St. Petersburg /ID# 256050, St. Petersburg, Florida
  - Southern Vitreoretinal Associates /ID# 256158, Tallahassee, Florida
  - Southeast Retina Center /ID# 256022, Augusta, Georgia
  - Georgia Retina - Marietta /ID# 256142, Marietta, Georgia
  - Marietta Eye Clinic /ID# 268163, Marietta, Georgia
  - Thomas Eye Group PC /ID# 268159, Sandy Springs, Georgia
  - Retina Consultants of Hawaii /ID# 256049, ‘Aiea, Hawaii
  - University of Illinois at Chicago /ID# 256300, Chicago, Illinois
  - University Retina and Macula Associates /ID# 256078, Lemont, Illinois
  - University Retina and Macula Associates /ID# 256077, Oak Forest, Illinois
  - Springfield Clinic /ID# 266225, Springfield, Illinois
  - Retina Partners Midwest, PC /ID# 256045, Indianapolis, Indiana
  - John-Kenyon American Eye Institute -New Albany /ID# 256065, New Albany, Indiana
  - Retina Associates - Lenexa /ID# 256080, Lenexa, Kansas
  - Cincinnati Eye Institute- Edgewood /ID# 256132, Edgewood, Kentucky
  - Retina Associates of New Orleans /ID# 272440, Metairie, Louisiana
  - Ochsner Medical Center - Jefferson Highway /ID# 270524, New Orleans, Louisiana
  - The Retina Care Center /ID# 256144, Baltimore, Maryland
  - Johns Hopkins Hospital /ID# 256015, Baltimore, Maryland
  - The Retina Group Of Washington - Chevy Chase /ID# 276039, Chevy Chase, Maryland
  - Cumberland Valley Retina Consultants - Hagerstown /ID# 256151, Hagerstown, Maryland
  - Ophthalmic Consultants of Boston /ID# 256014, Boston, Massachusetts
  - Retina Associates of Michigan /ID# 266198, Grand Blanc, Michigan
  - Associated Retinal Consultants /ID# 256156, Royal Oak, Michigan
  - VitreoRetinal Surgery PLLC DBA Retina Consultants of Minnesota /ID# 256160, Edina, Minnesota
  - Mayo Clinic - Minnesota /ID# 256051, Rochester, Minnesota
  - The Retina Institute /ID# 266587, St Louis, Missouri
  - Sierra Eye Associates /ID# 256020, Reno, Nevada
  - Eye Associates of New Mexico /ID# 256075, Albuquerque, New Mexico
  - Long Island Vitreoretinal Consultants /ID# 256074, Great Neck, New York
  - Retina-Vitreous Surgeons of Central New York - Liverpool /ID# 266274, Liverpool, New York
  - Duke Eye Center /ID# 256076, Durham, North Carolina
  - Atrium Health Wake Forest Baptist Medical Center /ID# 270767, Winston-Salem, North Carolina
  - Retina Associates of Cleveland-Middleburg Heights /ID# 256052, Cleveland, Ohio
  - Cleveland Clinic Main Campus /ID# 256064, Cleveland, Ohio
  - Retina Vitreous Center, Research /ID# 256067, Edmond, Oklahoma
  - Verum Research, LLC /ID# 266585, Eugene, Oregon
  - Retina Northwest, PC /ID# 256140, Portland, Oregon
  - Erie Retina Research /ID# 256154, Erie, Pennsylvania
  - Retina Vitreous Consultants - Monroeville /ID# 271654, Monroeville, Pennsylvania
  - Mid Atlantic Retina /ID# 256013, Philadelphia, Pennsylvania
  - Charleston Neuroscience Institute /ID# 256235, Ladson, South Carolina
  - Black Hills Regional Eye Institute /ID# 256161, Rapid City, South Dakota
  - Charles Retina Institute /ID# 256016, Germantown, Tennessee
  - Retina Research Institute of Texas /ID# 256141, Abilene, Texas
  - Austin Research Center for Retina /ID# 256148, Austin, Texas
  - Austin Retina Associates - Austin /ID# 256053, Austin, Texas
  - Austin Clinical Research, LLC /ID# 256043, Austin, Texas
  - Retina Consultants of Texas - Beaumont /ID# 266279, Beaumont, Texas
  - Retina and Vitreous of Texas /ID# 263961, Bellaire, Texas
  - Texas Retina Associates - Dallas /ID# 256133, Dallas, Texas
  - Baylor Scott & White Surgicare /ID# 256122, Fort Worth, Texas
  - Retina Consultants Of Texas /ID# 268611, San Antonio, Texas
  - Stone Oak Surgery Center /ID# 266199, San Antonio, Texas
  - Retina Center Of Texas (Rct) - Southlake /ID# 256056, Southlake, Texas
  - Retina Consultants - The Woodlands /ID# 256018, The Woodlands, Texas
  - Retina Associates of Utah /ID# 256044, Salt Lake City, Utah
  - John A. Moran Eye Center /ID# 256068, Salt Lake City, Utah
  - Wagner Macula & Retina Center - Norfolk /ID# 256134, Norfolk, Virginia
  - Pacific Northwest Retina /ID# 256155, Bellevue, Washington
  - Retina Center NW, PLLC /ID# 256157, Silverdale, Washington
  - University of Wisconsin-Madison, Department of Ophthalmology and Visual Sciences /ID# 256159, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=RGX-314-2104